CLINICAL TRIAL: NCT05084807
Title: Evaluation of the Lymphocyte Subpopulations in the Normal Mucosa of the Upper Digestive Tract
Acronym: GUTproject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GUT2020
Record Dates: First submitted 2021-09-28; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Lymphocytic Enteritis (Disorder); Healthy Volunteers
Keywords: Intraepithelial Lymphocytes; Intraepithelial T Cells; Celiac Disease; Crohn Disease; Healthy Volunteers
MeSH Terms: conditions — Celiac Disease; Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Study Type: descriptive cross-sectional study, prospective. Estimated enrollment: 20 individuals. Estimated duration of the project: 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy group (Other): A group of healthy, strictly asymptomatic individuals of both sexes and different age groups.
  Interventions: Other: Endoscopy

INTERVENTIONS:
Other: Endoscopy — * A dyspepsia test will be performed to avoid selection bias. In subjects strictly asymptomatic, a blood analysis will be proposed.
  * Subjects who present strictly normal laboratory tests (including celiac serology and negative H Pylori tests) and no genetic risk of celiac disease will be invited to perform an upper gastrointestinal endoscopy.
  * During gastroscopy, samples of normal mucosa will be taken for histological and lymphocyte subpopulations analysis. The percentage of lymphocyte subpopulations will be assessed by flow cytometry.
  * To compare whether there are differences between the lymphocyte subpopulations related to the age and sex of the healthy individuals, a student's t test, ANOVA or the corresponding non-parametric test will be used. The values will be expressed according to: mean +/- 2DS or median and interquartile range.

SUMMARY:
The macro and microscopic findings of the upper gastrointestinal tract are useful in the differential diagnosis of digestive diseases such as Crohn's or celiac diseases. However, the histopathological findings (duodenal lymphocytosis, atrophy, chronic inflammatory infiltrate, etc.) are generally not pathognomonic, and there is a great overlap between different inflammatory diseases. The study of lymphocyte subpopulations of the intestine has shown its usefulness in cases of celiac disease that are difficult to diagnose. In patients with celiac disease, lymphocytes that infiltrate the duodenum present a specific pattern with increased percentage of TCRgẟ+ lymphocytes and reduced percentage of CD3- lymphocytes. However, it is currently unknown if other inflammatory diseases (e.g. Crohn's disease) have specific lymphocyte subpopulations that could be of great diagnostic aid. One of the main problems in establishing patterns associated with disease is the absence of immunological studies carried out in healthy individuals. Most of the studies include, as a control group, patients who undergo gastroscopy for the study of upper digestive symptoms and have microscopically normal duodenal biopsy. This is a heterogeneous population that includes, among others, patients with functional pathology in whom the existence of low-grade inflammatory phenomena has been suggested. Therefore, patients with digestive symptoms are not good controls to establish normal patterns of intestinal immunity.

DETAILED DESCRIPTION:
Hypothesis: The evaluation of the lymphocyte subpopulations of the subjects without digestive symptoms and normal upper digestive tract mucosa will allow to have a healthy control group with which to compare the cellular patterns of different chronic inflammatory diseases.

ELIGIBILITY:
Study population: 20 healthy individuals, strictly asymptomatic, of both sexes, in different age groups will be included.

Inclusion Criteria:

* Adult individuals without any comorbidity, strictly asymptomatic.
* Age> 18 years.
* Informed consent signature.
* Carrying out a varied, non-restrictive diet.
* Negative blood tests including celiac serology, H. pylori serology and celiac disease genetic study (will only be accepted if they have positive DQ2.2 allele).
* Normal esophagogastroduodenoscopy.
* Grossly and microscopic normal duodenal mucosa.

Exclusion Criteria:

* Refusal of the individual to participate.
* Severe disease (heart disease, lung disease, liver disease, bleeding disorders, neoplasms, etc.).
* Personal history of celiac disease and / or inflammatory bowel disease.
* Pregnancy and/or lactation.
* Age> 45 years.
* BMI> 28.
* Presence of any current digestive symptoms (negative responses must be met in all items of the dyspepsia test).
* Family history of 1st or 2nd degree of celiac disease or inflammatory bowel disease.
* Potentially contagious diseases (HIV, HCV, HBV, tuberculosis, Covid19, ...).
* Trips to tropical countries in the last 6 months.
* Presence of coagulopathy or use of anticoagulant treatments.
* Consumption of any drug (including NSAIDs) in the last 4 weeks.
* Strict vegetarian, vegan or gluten-free diet.
* H. pylori positive.
* DQ2.5 positive and /or DQ8 positive
* Positive celiac serology (anti-transglutaminase> 2 U / mL).
* Active smoking.
* Habitual alcohol intake >40 g in men and 20 g in women.
* Alcohol intake in the previous 3 days.
* Esophagus-gastro-duodenoscopy with macroscopically abnormal mucosa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of the lymphocyte subpopulations of the upper digestive tract as assessed by flow cytometry in asymptomatic healthy subjects with normal mucosa. | 4 hour
  During gastroscopy, samples of normal mucosa will be taken for histological and lymphocyte subpopulations analysis. The percentage of lymphocyte subpopulations will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Comparison the percentage of the pattern of lymphocyte subpopulations in the duodenum in relation to age and sex. | 4 hour
  To compare whether there are differences between the lymphocyte subpopulations related to the age and sex of the healthy individuals, a student's t test, ANOVA or the corresponding non-parametric test will be used. The values will be expressed according to: mean +/- 2DS or median and interquartile range.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Esteve, PhD, MD, Principal Investigator — Hospital Universitari Mútua Terrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No